CLINICAL TRIAL: NCT02623543
Title: Effectiveness of Orthokeratology in Decreasing Myopic Progression in a Young Adult Population Enrolled in a Professional Optometric Curriculum
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illinois College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OK-ICO
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Myopia Progression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OrthoK (Experimental): OrthoK lenses will be prescribed for subjects randomly and followed for 2yrs throughout wearing the lenses. There will be an enrollment appointment, dispense appointment, 1-day, 1-week, 1-month, 6-month, 12-month, and 24-month follow-ups.
  Interventions: Device: OrthoK
- Control (Placebo Comparator): Subjects in the randomly assigned control will continue to wear their glasses throughout the 2yr follow-up period. There will be an enrollment appointment, 6-month, 12-month, and 24-month follow-ups.
  Interventions: Device: OrthoK

INTERVENTIONS:
Device: OrthoK

SUMMARY:
The high prevalence of myopia - especially in Asian countries - is well documented, as are the sight-threatening complications of high or degenerative myopia. Retinal detachment, glaucoma, vitreal degeneration and focal retinal changes occur secondary to the progressive axial elongation of the eye with age. Specialty rigid lenses have long been shown to lessen this progression in the pediatric population; orthokeratology (ortho-k) lenses are worn at night and change the corneal topography to correct low to moderate amounts of myopia. This same axial elongation has also been shown to occur in young adults with high near demands, however to our knowledge, there are no studies examining the effect of ortho-k lenses in this population. Our project seeks to investigate the efficacy of ortho-k in slowing axial elongation and myopic progression in subjects between the ages of 21-30. Results will help elucidate what role these specialty lenses may have in the management of the myopic patient throughout their development, as well as what potential they have in prevention of associated degenerative changes.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be in the incoming first year optometry class, with a myopic prescription between -0.50D and -5.00D in at least one eye with refractive astigmatism <1.50D. Visual acuity must be at least logMAR 0.10 (Snellen 20/25) or better at baseline examination in both eyes. Ocular examination must not reveal any strabismus, ocular pathology or contraindications for orthokeratology lens wear. Subjects must be in good general health with no systemic conditions that might impact their ocular health or refractive error. They must be willing to sleep a minimum of six hours per night. Finally, subjects must be willing and able to present to clinic for all necessary follow-up care.

Exclusion Criteria:

* Prescription falls outside the refractive guidelines, have a history of any type of trauma or ocular surgery, have a history of prior experience with myopia control treatment, are amblyopic or if they are current gas permeable lens wearers. They will be discontinued from the study if they are non-compliant with the treatment protocol or do not achieve a desirable subjective result,

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Myopia Progression | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States